CLINICAL TRIAL: NCT06510946
Title: Efficacy of an Intervention to Increase Therapeutic Adherence in Patients With Secondary Prevention for Cardiovascular Disease.
Brief Title: Improving Therapeutic Adherence in Cardiovascular Secondary Prevention.
Acronym: AT-PSC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Francisco Manuel Lidón Muñoz, Bachelor's in Medicine. PhD student., Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-016
Record Dates: First submitted 2024-07-13; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Chronic Disease; Secondary Prevention; Coronary Disease
Keywords: Treatment Adherence and Compliance; Primary Health Care
MeSH Terms: conditions — Cardiovascular Diseases; Chronic Disease; Coronary Disease; Treatment Adherence and Compliance | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: health education, use of mobile phones, personalized dosage system.
  Interventions: Behavioral: (Health education program) To increase therapeutic adherence in patients with secondary prevention for cardiovascular disease
- Control group (No Intervention): Routine follow-up.

INTERVENTIONS:
Behavioral: (Health education program) To increase therapeutic adherence in patients with secondary prevention for cardiovascular disease — The intervention involves a comprehensive health education program based on the Chronic Care Model to increase therapeutic adherence in patients with secondary prevention for cardiovascular disease. The program includes the following components:
  Health Education Sessions: Education on the importance of adherence, understanding the disease, side effects of medications, and their management. It addresses personal beliefs and concerns.
  Mobile Phone Reminders: Use of alarms and the ti.care® app to remind patients to take their medications.
  Medication Verification: Ensuring that the medications and dosages taken match the prescriptions.
  Personalized Dosing Systems (PDS): Helping manage medication intake.
  Additional Health Advice: Control of other cardiovascular risk factors and benefits of the Mediterranean diet.
  Arms: Intervention group

SUMMARY:
The goal of this open label randomized controlled trial is to evaluate the efficacy of an intervention through health education based on the Chronic Care Model's implementation to increase therapeutic adherence in patients with secondary prevention for cardiovascular disease. The main questions it aims to answer are:

* Null hypothesis (H0): In patients in cardiovascular secondary prevention, an intervention based on the application of the Chronic Care Model does not improve therapeutic adherence to the 3 preventive drugs: Angiotensin converting enzyme inhibitors/Angiotensin II receptor blockers, acetylsalicylic acid, and statins.
* Alternative hypothesis (H1): In patients in cardiovascular secondary prevention, an intervention based on the application of the Chronic Care Model improves therapeutic adherence to the 3 preventive drugs: Angiotensin converting enzyme inhibitors/Angiotensin II receptor blockers, acetylsalicylic acid, and statins.

Researchers will compare intervention group (health education, use of mobile phones, personalized dosage system) to the control group (routine follow-up).

DETAILED DESCRIPTION:
Cardiovascular diseases are the worldwide's leading cause of mortality. Within the spectrum of these diseases, cerebrovascular disease, coronary heart disease, and peripheral vascular disease are included. Secondary prevention is an effective strategy in patients with previous events, being the most used drugs antihypertensives, statins and salicylic acetyl acid.

Therapeutic adherence in these patients is crucial, as the lack of it, results in increased morbidity and mortality, as well as decreased quality of life and raised healthcare costs. However, less than half of the patients take all three medications during the first year. In addition, the lack of therapeutic adherence is easier to measure in the primary care setting.

Objective: To evaluate the efficacy of an intervention through health education based on the Chronic Care Model's implementation to increase therapeutic adherence in patients with secondary prevention for cardiovascular disease.

Methods: Open label randomized controlled trial, selecting patients presenting the inclusion criteria through consecutive probability sampling. Random assignment will be carried out using a random number table.

Intervention on patients in the experimental group will be conducted through health education following the recommendations of the Chronic Care Model (CCM). The aim is to empower patients to manage their disease through therapeutic education measures and shared decision-making with the patient.

Two individual sessions (one in the first month and another in the fourth month) and four group sessions (one per quarter with 5 to 10 patients) will be conducted. The individual sessions will last 30 minutes, and the group sessions will last 1 hour.

In the first quarter, an individual session will be held in the first month, followed by a group session in the second month. In the second quarter, another individual session will be held in the fourth month, and a group session in the sixth month. Subsequently, group sessions will continue with one scheduled in the ninth month and another in the twelfth month.

Considering a therapeutic adherence of 50% in the control group and an expected therapeutic adherence of 80% in the intervention group, with a type II error of 20% (80% power), a type I error of 5% (95% confidence interval), and a 15% loss rate, a sample size of 45 patients in each group is estimated.

The follow-up period will be conducted for one year. After data collection, a descriptive univariate analysis of the variables and a bivariate analysis will be performed. Finally, a multivariate analysis will be conducted to isolate potential confounding factors and to analyze the impact of the intervention on therapeutic adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged over 18 years old, who, after reading the patient information sheet, provide written informed consent.
* Patients in secondary prevention receiving daily single-dose angiotensin converting enzyme inhibitors/Angiotensin II receptor blockers, acetylsalicylic acid, and statins for 6 months or more.
* Diagnosis of any of the following cardiovascular diseases: cerebrovascular disease, ischemic heart disease, or peripheral vascular disease.
* Patients under follow-up at our primary care center.
* Patients identified with therapeutic adherence deficiency, defined as Haynes-Sackett test supplemented with Medication Possession Ratio (MPR) < 80% for any of the 3 drugs in the previous 6 months.

Exclusion Criteria:

* Patients who refuse to participate.
* Incomplete completion of informed consent.
* Language barrier.
* Patients diagnosed with psychiatric, psychological, neurological, and/or social problems that hinder intervention or follow-up.
* Life expectancy less than one year.
* Patients whose treatment is managed by a caregiver (professional or family member).
* Patients with Barthel Index <60.
* Institutionalized patients.
* Patients currently participating in similar research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic adherence | Through study completion, an average of 1 year.
  Its evaluation will be carried out using the Haynes-Sackett test to determine therapeutic adherence vs. non-adherence (dichotomous qualitative variable) complemented with the Medication Possession Ratio (MPR), estimating a percentage (continuous quantitative variable). Good adherence is considered if the patient reports no difficulties in taking all their pills and has an MPR > 80% for the 3 preventive drugs. Otherwise, it is considered poor therapeutic adherence. Poor therapeutic adherence is defined by the MPR if 20% or more of the prescribed packages have not been collected from the pharmacy in the last year. Poor adherence is determined if it is diagnosed by either method. As 3 drugs are analyzed, poor therapeutic adherence is considered if it occurs with any one of them, with two, or with all three.
  To evaluate therapeutic adherence, the Haynes-Sackett test will be administered, complemented by the MPR from the medical records.

SECONDARY OUTCOMES:
Group | This variable will be collected prior to the start of the study.
  Intervention group and control group
Age | This variable will be collected prior to the start of the study.
  Years old
Sex | This variable will be collected prior to the start of the study.
  Man and woman
Race | This variable will be collected prior to the start of the study.
  Caucasian Black Asian Hispanic Other
Educational level | This variable will be collected prior to the start of the study.
  Illiterate. Primary education (Elementary school or Compulsory Secondary Education). Vocational training and vocational education. High school diploma (Baccalaureate). Higher education: bachelor's degree, master's degree, and/or doctorate.
The Barthel index | This variable will be collected prior to the start of the study.
  The main aim is to establish degree of independence.
Quality of life studied using the European Quality of Life-5 Dimensions | This variable will be collected prior to the start of the study.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Manuel Lidón Muñoz, Principal Investigator — Universidad Miguel Hernández de Elche
Locations (1):
- Babel Health Centre, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lidon-Munoz FM, Quesada JA, Gil-Guillen VF, Orozco-Beltran D. Efficacy of an intervention to increase therapeutic adherence in patients with secondary prevention for cardiovascular disease: a study protocol for a randomized controlled trial. Front Med (Lausanne). 2025 Jan 7;11:1510744. doi: 10.3389/fmed.2024.1510744. eCollection 2024. PMID 39839644